CLINICAL TRIAL: NCT00199745
Title: Investigations on Differences in Atorvastatin Metabolite Ratios as a Diagnostic Tool in Detecting Atorvastatin Induced Myotoxicity
Brief Title: Differences in Atorvastatin Metabolite Ratios as a Diagnostic Tool in Detecting Atorvastatin Induced Myotoxicity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo School of Pharmacy (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Muskelbiopsistudie Lipid05-06; S-05229 (REK - Sør); 13041 (NSD)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Muscular Diseases
Keywords: statin; statins; statin therapy; adverse events; side effect; Myotoxicity; atorvastatin; Atorvastatin Therapy
MeSH Terms: conditions — Muscular Diseases; Myotoxicity | interventions — Atorvastatin

INTERVENTIONS:
Drug: atorvastatin

SUMMARY:
The primary objective of the study is to investigate whether differences in atorvastatin metabolite ratios might have a positive or negative predictive value in diagnosing atorvastatin muscle toxicity. A muscle biopsy is also collected and investigated.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate whether differences in atorvastatin metabolites ratios might have a positive or negative predictive value in diagnosing atorvastatin muscle toxicity. A muscle biopsy is also collected and investigated.

ELIGIBILITY:
Inclusion Criteria:

* Suspected atorvastatin induced muscle adverse events
* Signed informed consent
* 18 years of age or older
* Able to donate blood samples
* Ongoing treatment with atorvastatin (not necessary if patients only donate a muscle biopsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To compare ratios atorvastatin metabolites to atorvastatin in patients with confirmed atorvastatin-induced myopathy compared to healthy volunteers

SECONDARY OUTCOMES:
Phenotypic differences in isolated muscle cells of patients experiencing muscle toxicity compared to a control group

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Retterstøl, MD, Principal Investigator — Lipidklinikken, Rikshospitalet-Radiumhospitalet HF; Anders Åsberg, Associate Professor, Principal Investigator — Department of Pharmaceutical Biosciences, School of Pharmacy, University of Oslo
Locations (1):
- Lipidklinikken, Rikshospitalet-Radiumhospitalet HF, Oslo, Oslo County, Norway